CLINICAL TRIAL: NCT00084630
Title: A Phase II Study of Imatinib (NSC-716051) in Patients With Locally Advanced or Metastatic Dermatofibrosarcoma Protuberans
Brief Title: Imatinib Mesylate in Treating Patients With Locally Recurrent or Metastatic Dermatofibrosarcoma Protuberans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03184; S0345; U10CA032102 (NIH); CDR0000365465 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Adult Fibrosarcoma; Dermatofibrosarcoma Protuberans; Recurrent Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Fibrosarcoma; Dermatofibrosarcoma; Sarcoma | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once daily on days 1-56. Treatment repeats every 56 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with documented tumor progression and no serious side effects may continue therapy at a higher dose for another 6 courses.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well imatinib mesylate works in treating patients with locally recurrent or metastatic dermatofibrosarcoma protuberans (DFSP) or transformed fibrosarcomatous DFSP (a type of soft tissue sarcoma). Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate (confirmed complete and confirmed partial response) in patients with locally advanced or metastatic dermatofibrosarcoma protuberans (DFSP) treated with imatinib.

II. To estimate the one-year progression-free survival probability in this population when treated with imatinib.

III. To evaluate the frequency and severity of toxicities associated with this treatment.

IV. To measure the presence of PDGFB gene rearrangement in DFSP detectable by RT-PCR (for COL1A1-PDGFB fusions) and/or FISH (PDGFB rearrangements with unknown partners) and explore relationships between these measures and survival and tumor response in a preliminary manner.

V. To investigate in a preliminary fashion the correlation of plasma levels of imatinib after 1 month of treatment with the response of DFSP.

VI. To obtain tumor material for additional future correlative studies of the activity of intracellular kinases, cDNA microarray analyses and PDGFB receptor gene sequence analyses.

OUTLINE:

Patients receive oral imatinib mesylate once daily on days 1-56. Treatment repeats every 56 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with documented tumor progression and no serious side effects may continue therapy at a higher dose for another 6 courses.

Patients are followed every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of either dermatofibrosarcoma protuberans (DFSP) or transformed fibrosarcomatous DFSP; patients with transformed fibrosarcomatous DFSP may have primary, locally recurrent or metastatic disease; patients with DFSP must have locally recurrent or metastatic disease OR primary disease for which complete excision with a wide margin (> 1-2 cm) would result in unacceptable cosmetic disfigurement or functional impairment
* Patients must have measurable disease; x-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; x-rays, scans or other tests for assessment of non-measurable disease must have been performed within 42 days prior to registration; all disease must be assessed
* Pathology materials must be submitted for review; failure to submit pathology materials will render the patient ineligible
* Patients must be willing to have blood samples submitted for testing of drug levels; also, it is strongly recommended that patients submit fresh/frozen tumor tissue that will yield 0.5 grams (0.5 cubic centimeters) for molecular correlative studies related to the PDGFR pathway
* Patient must not have had chemotherapy, biologic therapy or investigational agents for this tumor within 28 days prior to registration
* Patients may have received prior major surgery for this disease; at least 14 days must have elapsed since the surgery and the patient must have recovered from all side effects associated with surgery; biopsy of dermatofibrosarcoma protuberans is not considered major surgery and a 14-day delay after biopsy is not required
* Prior radiotherapy is allowed, provided at least four weeks have elapsed since the last treatment, there is evidence of progressive disease within or measurable disease outside of the radiation field, and the patient must have recovered from all associated toxicities at the time of registration
* Patients must have Zubrod performance status of =< 2
* WBC >= 2,000/uL
* ANC >= 1,500/uL
* Platelets >= 100,000/uL
* Serum bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Serum transaminase (SGOT or SGPT) must be =< 2.5 x IULN
* Serum albumin must be >= 2.5 mg/dl
* Patients must not be taking therapeutic doses of coumadin (Warfarin) at the time of registration; patients requiring therapeutic anticoagulation may use heparin, low molecular weight heparin or other agents; mini-dose coumadin (1 mg orally every day as prophylaxis is allowed
* Patients with known CNS metastases are not eligible
* Pregnant or nursing women may not participate on this study; there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with imatinib; male/female patients of reproductive potential must also agree to employ an effective contraceptive barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patients registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study have been entered into the database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Response rate (confirmed complete and confirmed partial response) | Up to 5 years
Progression-free survival | At 1 year
Frequency and severity of toxicity as assessed by NCI CTCAE version 3.0 | Up to 5 years after completion of treatment
Relationship between PDGFB and survival | At baseline and at the time of progression

SECONDARY OUTCOMES:
Relationship between PDGFB and tumor response to imatinib mesylate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States